CLINICAL TRIAL: NCT03284398
Title: Observational Retrospective Analysis Assessing the Influence of Three-Chamber Bags Compared to Hospital Compounded Parenteral Nutrition Bags on Blood Stream Infections
Brief Title: Three-Chamber Bags Retrospective Study in Spain
Status: Completed | Type: Observational
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Other Study IDs: 3CBs-001-CNI
Record Dates: First submitted 2017-09-04; First posted 2017-09-15 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Parenteral Nutrition; Blood Stream Infection
Keywords: parenteral nutrition; ICU; 3-chamber bags; ICD-9-CM; BSI; Medical records system; computerized
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parenteral nutrition bag type: Groups with different parenteral nutrition bags (3CBs or HCBs)

SUMMARY:
The primary study objective is to assess the rates of blood stream infection (BSI) from the use of Three-Chamber Bags (e.g., SmofKabiven®, Kabiven®, others) compared to Hospital Compounded Bags (HCBs) in patients requiring parenteral nutrition in Spanish hospitals.

DETAILED DESCRIPTION:
This is a retrospective observational database study of patients receiving parenteral nutrition (PN) for at least 3 consecutive days with hospital admission date between January 1, 2013, and December 31, 2015 (study period).

The study will use an as treated approach, where patients will be followed from the index date (hospital admission day of the hospitalization during which PN is administered) up to patient discharge or death (observation period).

The study will be conducted using an initial EMR (Electronic Medical Record) data retrieval process, followed by manual data retrieval (chart review) that will complement data obtained from EMR. Data collection for manual data retrieval will be conducted through an eCRF.

The documentation of patient data will comprise two sequential steps. The initial step will include data of 30% of patients and then an interim analysis (IA) will be conducted. If IA shows positive results, data for the remaining 70% of patients (step II) will be gathered.

The study will be conducted in 10-14 sites in Spain.

Data analysis: Baseline demographics, co-morbidities, and hospitalization characteristics will be reported descriptively by means of mean with standard deviations and medians with ranges for continuous variables and by counts and percentages for categorical variables. Incidence rates for BSI will be reported by treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Adult hospital inpatients ≥ 18 years
2. Treatment with PN for at least 3 consecutive days
3. PN containing all three major macronutrients, delivered from 3CB or HCB
4. Patients with hospital admission between January 1, 2013, and December 31, 2015 (study period)

Exclusion Criteria:

1. Bloodstream infection before or at the same day of first PN administration
2. Immunosuppression due to concomitant therapy (e.g., immunosuppressive therapy due to transplantation, concomitant oral or intravenous administration of glucocorticoids) or disease (e.g., HIV, leukaemia)
3. Permanent vascular access (port, shunts for dialysis)
4. Femoral venous placement of central venous line used for PN
5. Burns, extensive skin injuries (e.g., Lyell´s disease)
6. Chemo-/radiotherapy for up to 3 months before hospital admission
7. Change of PN bag type during observation period, e.g., from HCBs to 3CBs or vice-versa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Population will include adult hospitalized patients receiving PN, treated on any ward and by any medical discipline within the hospital (e.g., intensive care unit, normal wards; surgery, non-surgery) during the study period. For every patient, one hospitalization episode will be documented.
Sampling Method: Probability Sample
Enrollment: 3723 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Stover, Study Chair — Fresenius Kabi Deutschland GmbH, Borkenberg 14, 61440 Oberursel, Germany; Juan Carlos M González, Principal Investigator — Hospital Universitario 12 de Octubre, 28041 Madrid, Spain
Locations (2):
- Spain (2):
  - Hospital de Manacor, Manacor, Balearic Islands
  - Hospital Universitario 12 de Octubre, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective cohort study. Data collection from medical records
Groups:
- Three-chambered Bag (3CB): Hospitalized adults (≥18 years) who received PN containing all three major macronutrients via an industrially-compounded three-chambered PN bag for ≥3 consecutive days during the study period
- Hospital-Compounded Bag (HCB): Hospitalized adults (≥18 years) who received PN containing all three major macronutrients via a Hospital-compounded all-in-one PN bag for ≥3 consecutive days during the study period
Period: Overall Study
Arm/Group | Three-chambered Bag (3CB) | Hospital-Compounded Bag (HCB)
Started | 2753 | 970
Completed (Retrospective data collection: all patients under study intervention during the predefined period) | 2753 | 970
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 5389 patient records were screened for eligibility; of these, 3723 met the selection criteria, including 2753 patients who received 3CB and 970 patients who received MCB
Groups:
- Three-Chambered Bag (3CB): Hospitalized adults (≥18 years) who received PN containing all three major macronutrients via industrially-compounded 3CB for ≥3 consecutive days during the observation period (January 1, 2013 to December 31, 2015).
- Hospital-compounded Bag (HCB): Hospitalized adults (≥18 years) who received PN containing all three major macronutrients via hospital-compounded all-in-one bag for ≥3 consecutive days during the observation period (January 1, 2013 to December 31, 2015).
- Total: Total of all reporting groups
Arm/Group | Three-Chambered Bag (3CB) | Hospital-compounded Bag (HCB) | Total
Number analyzed (Participants) | 2753 | 970 | 3723
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (15.2) | 66.5 (14.8) | 66.8 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1144 | 354 | 1498
  Male | 1609 | 616 | 2225
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 2753 | 970 | 3723

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Presenting With a Confirmed Microbial Blood Stream Infection During Treatment With PN for Each Group (3CB vs HCB)
Description: Confirmation of BSI required fulfillment of all of the following criteria:
  * International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9-CM) code for sepsis (038.x), septicemia (995.91), severe sepsis (995.92), septic shock (785.52), bacteremia (790.7), unspecified infection due to central venous catheter (999.31), or BSI due to central venous catheter (999.32)
  * Positive blood culture collected during PN administration
  * Concomitant antimicrobial therapy
Time Frame: Entire study period, from January 1, 2013 and December 31, 2015
Measure: Count of Participants; unit: Participants
Groups:
- Three-Chambered Bag: Treatment with industrially-compounded PN formulation in three-chambered bag
- Hospital-compounded Bag: Treatment with Hospital-compounded PN bag
Arm/Group | Three-Chambered Bag | Hospital-compounded Bag
Number analyzed (Participants) | 2753 | 970
Participants | 127 | 106

2. Secondary Outcome: Sepsis During PN
Description: Percentage of patients presenting at least one episode of Sepsis during treatment with PN for each group (3CB vs HCB)
Time Frame: From date of admission to date of discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Three-Chambered Bag (3CB) | Hospital-Compounded Bag (HCB)
Number analyzed (Participants) | 2753 | 970
Participants | 431 | 228

3. Secondary Outcome: Treatment With Antimicrobials During PN
Description: Percentage of patients receiving antimicrobial agents during treatment with PN for each group (3CB vs HCB)
Time Frame: Any day during PN treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Three-chambered Bag (3CB) | Hospital-Compounded Bag (HCB)
Number analyzed (Participants) | 2753 | 970
Participants | 831 | 370

4. Secondary Outcome: Use of Vasopressor Treatment
Description: Percentages of patients requiring vasopressor support during PN treatment
Time Frame: Patients requiring vasopressor support at any time during treatment with PN
Measure: Count of Participants; unit: Participants
Arm/Group | Three-Chambered Bag (3CB) | Hospital-compounded Bag (HCB)
Number analyzed (Participants) | 2753 | 970
Participants | 410 | 291

5. Secondary Outcome: Use of Mechanical Ventilation
Description: Percentage of patients requiring mechanical ventilation during PN treatment for each group (3CB vs HCB)
Time Frame: Patients requiring mechanical ventilation at any time during PN treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Three-Chambered Bag (3CB) | Hospital-compounded Bag (HCB)
Number analyzed (Participants) | 2753 | 970
Participants | 410 | 299

6. Secondary Outcome: Renal Replacement Therapy
Description: Percentage of patients requiring Renal Replacement Therapy during PN treatment for each group (3CB vs HCB)
Time Frame: Patients requiring renal replacement therapy for at least one day during PN treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Three-Chambered Bag (3CB) | Hospital-compounded Bag (HCB)
Number analyzed (Participants) | 2753 | 970
Participants | 78 | 89

7. Secondary Outcome: Newly-occurred Abnormal Laboratory Findings During PN
Description: Percentage of patients presenting newly-occurred abnormal laboratory results during PN for each group (3CB vs HCB)
Time Frame: During PN treatment inclusive day 1
Population: Simultaneous occurring laboratory abnormalities
Measure: Count of Participants; unit: Participants
Arm/Group | Three-Chambered Bag (3CB) | Hospital-compounded Bag (HCB)
Number analyzed (Participants) | 2753 | 970
Participants
  Metabolic impairment | 1193 | 584
  Any hepatic dysfunction | 1414 | 651
  Any abnormal electrolytes | 1444 | 699

8. Secondary Outcome: Organ Failure
Description: Percentage of patients presenting at least one organ failure during treatment with PN for each group (3CB vs HCB)
Time Frame: Any time during PN treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Three-Chambered Bag (3CB) | Hospital-compounded Bag (HCB)
Number analyzed (Participants) | 2753 | 970
Participants
  Any organ failure | 905 | 562
  Single organ failure | 593 | 255
  Multiple organ failure | 312 | 307

9. Secondary Outcome: Hospital Length of Stay (LOS)
Description: Hospital length of stay in days for patients for each group (3CB vs HCB)
Time Frame: Duration in days from admission to death or discharge for each treatment arm
Measure: Number; unit: Days
Arm/Group | Three-Chambered Bag (3CB) | Hospital-compounded Bag (HCB)
Number analyzed (Participants) | 2753 | 970
Days | 26,601 | 30,384

10. Secondary Outcome: Length of Stay in the ICU
Description: Total number of days in the ICU for each group (3CB vs HCB)
Time Frame: All patients admitted in the ICU at any time during PN treatment
Measure: Number; unit: Days
Arm/Group | Three-Chambered Bag (3CB) | Hospital-compounded Bag (HCB)
Number analyzed (Participants) | 2753 | 970
Days | 3,017 | 3,772

ADVERSE EVENTS:
Time Frame: Retrospective, observational, non-interventional study. All-cause mortality, Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: Not applicable since study was retrospective, observational/non-interventional. All-cause mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Groups:
- Three-Chambered Bag (3CB); Hospital-compounded Bag (HCB): Not applicable (Observational/non-interventional retrospective data collection)
Arm/Group | Three-Chambered Bag (3CB) | Hospital-compounded Bag (HCB)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03284398/Prot_SAP_000.pdf